CLINICAL TRIAL: NCT06222840
Title: Electro-clinical Features and Functional Connectivity Analysis in SYN1 Gene Mutation-related Epilepsy
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN662023/CHUSTE
Record Dates: First submitted 2023-12-12; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-07

CONDITIONS: Epileptic Syndromes
Keywords: SYN1 mutation; reflex bathing epilepsy; neurodevelopmental disorders; connectivity analysis; electro-encephalographic seizure pattern
MeSH Terms: conditions — Epileptic Syndromes; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: cases with SYN1 gene mutation
  Interventions: Other: Electro-clinical analysis of epileptic seizures; Other: Electro-encephalographic cases; Other: Clinical datas analysis
- Arm 2: control cases
  Interventions: Other: Electro-encephalographic control

INTERVENTIONS:
Other: Electro-clinical analysis of epileptic seizures — Electro-clinical analysis of epileptic seizures
  Groups: Arm 1
Other: Electro-encephalographic cases — Electro-encephalographic connectivity analysis compared to controls
  Groups: Arm 1
Other: Clinical datas analysis — Clinical datas analysis
  Groups: Arm 1
Other: Electro-encephalographic control — Electro-encephalographic connectivity analysis compared to cases
  Groups: Arm 2

SUMMARY:
SYN1 gene mutation is an X-linked gene mutation that causes numerous pathological manifestations such as seizures and neurodevelopmental disorders. A few descriptions of this disease have been published in the last decade, but the electro-clinical features of epilepsy are still largely unknown. No analysis of electroencephalographic connectivity has yet been performed. The aim of this study is to perform a detailed electro-clinical seizure analysis and electroencephalographic analysis in patients with a SYN1 gene mutation, in an attempt to identify a characteristic pattern that would allow earlier diagnosis and better understanding and management of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Cases : SYN1 gene mutation, available electroencephalographic and clinical data.
* Controls : older than 12 years at the moment of the electroencephalogram recording, electroencephalogram considered as normal, no neurological disease (particularly no epilepsy), no neuroimaging abnormality.

Exclusion Criteria:

- Controls : younger than 12 years at the moment of the electroencephalogram recording, electroencephalogram considered as abnormal, neurological disease (particularly epilepsy), neuroimaging abnormality.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SYN1 gene mutation patients and controls
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Electroencephalographic functional connectivity mapping | Month 6
  Identify a characteristic electroclinical pattern in SYN1 gene mutation related epilepsy

SECONDARY OUTCOMES:
Electroencephalographic reading grid | Month 6
  Compare electro-encephalographic connectivity between SYN1 gene mutation patients and controls

CONTACTS AND LOCATIONS:
Overall Officials: Laure MAZZOLA, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No